CLINICAL TRIAL: NCT03638063
Title: Adenosine Triphosphate and Capsaicin Cough Provocation Test for Identifing Patients With Chronic Cough Who Have Differential Responses to Purinergic Receptor Antagonists: a Randomized, Cross-over, Single-blind Trial
Brief Title: ATP and Capsaicin Cough Provocation Test in Chronic Cough and Bronchiectasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weijie Guan, Associated professor; principal investigator (respiratory medicine), Guangzhou Institute of Respiratory Disease
Other Study IDs: GuangzhouIRD01
Record Dates: First submitted 2018-08-13; First posted 2018-08-20 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Chronic Cough; Bronchiectasis
Keywords: Adenosine triphosphate; Capsaicin; cough provocation test
MeSH Terms: conditions — Chronic Cough; Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chronic cough: patients with chronic cough who remain clinically stable
  Interventions: Diagnostic Test: Adenosine Triphosphate; Diagnostic Test: capsaicin
- Bx: bronchiectasis patients who remain clinically stable
  Interventions: Diagnostic Test: Adenosine Triphosphate; Diagnostic Test: capsaicin
- Control: healthy controls
  Interventions: Diagnostic Test: Adenosine Triphosphate; Diagnostic Test: capsaicin

INTERVENTIONS:
Diagnostic Test: Adenosine Triphosphate — Adenosine Triphosphate aerosol
Diagnostic Test: capsaicin — capsaicin aerosol

SUMMARY:
This is a randomized, cross-over, single-blind trial. Eligible patients will be randomly assigned to undergo either capsaicin or adenosine triphosphate (ATP) cough provocation test, followed by a washout period of 2 to 14 days. Participants will be crossed-over to undergo another cough provocation test. Patient would be under observation in the out-patient clinics for ~2 hours following the cough provocation tests in case of severe adverse events.

DETAILED DESCRIPTION:
This is a randomized, cross-over, single-blind trial. After verification of the entry criteria, eligible patients will be, based on the randomization codes, randomly assigned to undergo either capsaicin or ATP cough provocation test (the participants will inhale capasaicin or ATP incremental concentration to induce cough, meanwhile the number of coughs and adverse events will be recorded in each concentration during the first 30 seconds), followed by a washout period of 2 to 14 days (no major changes in the use of concomitant medications are allowed,especially the medcines which are not allowed before test ). Participants will be crossed-over to undergo another cough provocation test. Patient would be under observation in the out-patient clinics for ~2 hours following the cough provocation tests in case of severe adverse events. Twenty four hours after each test, a follow-up telephone visit will be scheduled for all patients to record any response which may be related to the test.

ELIGIBILITY:
Inclusion Criteria:

* Out-patients of either gender, ex- or never-smokers, aged between 18 and 60 years
* Cough symptoms lasting for more than 8 weeks
* Remaining free of acute upper respiratory tract infection for at least 4 weeks
* Agreed to participate in the trial and signed informed consent.

Exclusion Criteria:

* Patients with serious systemic diseases (such as malignant tumors), bullae, severe uncontrolled asthma, and a history of major hemoptysis
* Systemic antibiotic use (except for maintenance low-dose macrolides) within 4 weeks
* Pregnancy or lactation
* Any known history of sensitivity to ATP or capsaicin
* Poor understanding of the test procedure
* Diagnosed with cough variant asthma or Eosinophilic bronchitis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patients with chronic cough (including bronchiectasis) who remained clinically stable for at least 4 weeks
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
C5 (Provocant concentration eliciting at least 5 coughs) | 18 months
  Provocant concentration eliciting at least 5 coughs

SECONDARY OUTCOMES:
ED50 (half maximal effective Dose) | 18 months
  50% effective dose of provocant
Emax (effective concentration of provocant eliciting maximal cough count) | 18 months
  effective concentration of provocant eliciting maximal cough count
potency ratio | 18 months
  ATP/capsaicin potency ratio
Difference in cough VAS score (a 10-point likert scale for assessing the global severity of cough, no subscale was applied) | 18 months
  The difference between pre- and post-challenge cough VAS scores
The incidence of adverse events (i.e. dry throat , pharyngeal itching) | 18 months
  adverse events such as dry throat , pharyngeal itching, wheeze or dyspnea according to the subject's reporting to record the rate of the incidence and the severity (the aboved-mentioned VAS score would be applied)
Cough dose ratio (CDR) | 18 months
  the ratio of cough count and dose/concentration

CONTACTS AND LOCATIONS:
Overall Officials: Ke-fang Lai, MD, Study Chair — Guangzhou Institute of Respiratory Health Locations: China, Guangdong First Affiliated Hospital of Guangzhou Medical
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Fowles HE, Rowland T, Wright C, Morice A. Tussive challenge with ATP and AMP: does it reveal cough hypersensitivity? Eur Respir J. 2017 Feb 8;49(2):1601452. doi: 10.1183/13993003.01452-2016. Print 2017 Feb. PMID 28179439
- [Background] Guan WJ, Gao YH, Xu G, Lin ZY, Tang Y, Li HM, Lin ZM, Zheng JP, Chen RC, Zhong NS. Capsaicin cough sensitivity and the association with clinical parameters in bronchiectasis. PLoS One. 2014 Nov 19;9(11):e113057. doi: 10.1371/journal.pone.0113057. eCollection 2014. PMID 25409316
- [Background] Torrego A, Haque RA, Nguyen LT, Hew M, Carr DH, Wilson R, Chung KF. Capsaicin cough sensitivity in bronchiectasis. Thorax. 2006 Aug;61(8):706-9. doi: 10.1136/thx.2005.049767. Epub 2006 Apr 6. PMID 16601085
- [Background] Fuller RW. Cough provocation tests: their clinical value. Pulm Pharmacol Ther. 2002;15(3):273-6. doi: 10.1006/pupt.2002.0355. PMID 12099777